CLINICAL TRIAL: NCT01219686
Title: Antidepressant Effect of Escitalopram: Delay of Onset. Clinical Randomized Double-blinded Study With Three Parallel Treatment Groups (Escitalopram 20mg vs Escitalopram 30mg vs Escitalopram 20 mg + Pindolol 15 mg/Day
Brief Title: EScitalopram PIndolol ONset of Action
Acronym: ESPION
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Markus KOSEL (Other)
Collaborators: University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); University Hospital, Basel, Switzerland (Other); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor-Investigator, Markus KOSEL, MD-PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 09-054, Psy 09-004
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Unipolar Depression
Keywords: unipolar depression, escitalopram, pindolol
MeSH Terms: conditions — Depressive Disorder | interventions — Escitalopram; Pindolol; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- escitalopram 20mg + pindolol 15mg (Experimental): Days 1-2: escitalopram 10 mg + placebo, days 3-42: escitalopram 20mg + placebo Days 1-14: pindolol 15 mg, days 15-17: pindolol 7.5 mg
  Interventions: Drug: escitalopram, pindolol
- Escitalopram 30 mg (Active Comparator): Days 1-2: escitalopram 10 mg+ placebo, days 3-4 escitalopram 20 mg + placebo, days 5-42: escitalopram 30mg+ placebo
  Interventions: Drug: escitalopram
- escitalopram 20 mg (Active Comparator): days 1-2: escitalopram 10 mg+ placebo, days 3-42: escitalopram 20 mg + placebo
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram, pindolol — escitalopram p.o., once daily, day 1-2: 10mg, days 3-42: 20mg pindolol p.o., twice daily 7.5 mg days 1-14, once daily 7.5 mg days 15-17
  Other Names: escitalopram/Cipralex; pindolol/Viskene
  Arms: escitalopram 20mg + pindolol 15mg
Drug: escitalopram — escitalopram p.o., once daily. days 1-2: 10 mg, days 3-4: 20 mg, days 5-42: 30 mg
  Arms: Escitalopram 30 mg
Drug: escitalopram — escitalopram 20 mg, p.o., once daily. Days 1-2: 10mg, days 3-42: 20 mg
  Arms: escitalopram 20 mg

SUMMARY:
The main purpose of this study is to determine whether the antidepressant response of escitalopram 30mg/day or escitalopram 20mg/day + pindolol, a beta blocker, is different (faster) compared to a standard dose of escitalopram 20mg/day.

DETAILED DESCRIPTION:
Antidepressant drug therapy is the primary therapeutic treatment option in moderate to severe Major Depressive Disorder. However, clinically significant antidepressant response needs sustained treatment during weeks to months. Indeed, in the largest effectiveness study conducted to date (STAR*D study) involving nearly 3000 depressed outpatients, only about one third of those who ultimately responded did so after 6 weeks of drug treatment and for most patients longer treatment periods were necessary. This delay implies prolonged suffering for the patients and their families. By its antagonist action on the serotonin 1A receptor pindolol is hypothesized to reduce the down-regulation mechanisms of antidepressants. It is therefore expected that addition of pindolol to escitalopram will shorten the therapeutic response. Clinical and preclinical data indicate that escitalopram at 30 mg/day might be more effective and perhaps be associated with a faster onset of action than 20mg. For this purpose the speed of action will be compared between three blindly randomized samples:

* escitalopram 20mg per day + placebo
* escitalopram 30mg per day + placebo
* escitalopram 20mg per day + pindolol 15mg per day (two doses of 7.5mg during 14 days).

Subjects will be followed for 6 weeks. The dose of 15mg pindolol per day (during 14 days) is based on the optimal occupancy of the serotonin 1A receptor.

At inclusion all subjects will be assessed by a trained psychiatrist using the SCID I mood disorder part which is based on DSM IV criteria, and by means of the French version of the MINI. Severity of depression will be assessed using the MADRS clinician rated and self-report questionnaire, and the French version of the QIDS.

Each week subjects will be assessed using the two versions of the Montgomery-Asberg Depression Rating Scale (MADRS) and the HCL-32 a self-report questionnaire assessing hypomania.

It is planned to include 135 patients during the three years of the study duration resulting in 45 subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65 years old
* patients suffering from major depression according to DSM-IV with a MADRS score of at least 25 and not treated by an antidepressant at the time of inclusion with the exception of non-responders to antidepressant for a period of at least 6 weeks or not tolerating an ongoing antidepressant necessitating a change of the antidepressant(excluding fluoxetine and irreversible MAOI)
* informed consent

Exclusion criteria:

* any other Axis I disorder excluding anxiety disorder not dominating the clinical picture, nicotine abuse
* non-responders to escitalopram in the past
* already taking pindolol
* pregnancy and breast feeding
* contraindication to one of the two treatments (medical conditions, drug treatments)
* significant somatic comorbidity interfering with the study procedures
* high risk of suicidality
* women of childbearing age not having a safe means of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
MADRS score change between baseline and 2 weeks of treatment | day 14
  Differences in MADRS score changes (baseline-day 14) between treatment groups

SECONDARY OUTCOMES:
Response/remission (MADRS) at 6 weeks | day 42
  % of patients with a given treatment which meet response/remssion criteria after 6 weeks of treatment, based on MADRS
Adverse events | See primary outcome measure
  Frequence of adverse events in treatment groups
Correlation of drug level of pindolol and/or escitalopram and clinical outcome (primary outcome) between treatment groups | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kosel, MD-PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Centre de Thérapies Breves (CTB), Secteur Jonction, Geneva, Switzerland